CLINICAL TRIAL: NCT00004487
Title: Phase III Study of Chondrocyte Alginate Gel Suspension in Pediatric Patients With Vesicoureteral Reflux
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Curis, Inc. (Industry)
Purpose: Treatment
Other Study IDs: 199/14267; REPRO-FDR001514; REPRO-99-07
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-04

CONDITIONS: Vesicoureteral Reflux
Keywords: rare disease; renal and genitourinary disorders; vesicoureteral reflux
MeSH Terms: conditions — Vesico-Ureteral Reflux; Rare Diseases; Urogenital Diseases

INTERVENTIONS:
Drug: chondrocyte-alginate gel suspension

SUMMARY:
OBJECTIVES: I. Determine the safety and efficacy of chondrocyte alginate gel suspension in pediatric patients with vesicoureteral reflux.

II. Determine the long term efficacy of this treatment regimen in this patient population.

III. Evaluate the short and long term avoidance of surgery or antibiotic therapy after this treatment regimen in this patient population.

IV. Estimate the risk:benefit ratio of this treatment regimen in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a multicenter study. Patients undergo biopsy of the auricular cartilage for chondrocytes during cystoscopic evaluation on day 1. Chondrocyte alginate gel suspension is injected into the submucosa of the bladder at the vesicoureteral junction between days 40-50. Patients found to have post treatment reflux may be retreated once.

Patients are followed at 1, 3, and 12 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Confirmed grade 3 or 4 reflux in at least one ureter by voiding cystourethrogram Breakthrough urinary tract infection despite standard antibiotic therapy OR Persistent reflux unlikely to resolve spontaneously
* Grade 3: 2 year reflux duration OR 1 breakthrough infection Grade 4: 1 year reflux duration OR 1 breakthrough infection
* Coexisting grade 1 or 2 reflux OR Resolved reflux (i.e., contralateral to the existing grade 3 or 4 refluxing ureter) allowed
* No reflux secondary to obstruction or neuropathic disease
* No gross urological abnormalities (e.g., megaureter requiring ureteral tapering or duplicity of ureters)

--Prior/Concurrent Therapy--

* Surgery: No prior surgery for correction of reflux No recent prior urological device implantation

--Patient Characteristics--

* Hematopoietic: No history of bleeding disorders
* Cardiovascular: No history of hypertension or cardiac disease
* Pulmonary: No history of pulmonary disease
* Other: No known allergies to contrast dyes, iodine, or shellfish No contraindications to general anesthesia No prior infections (other than UTIs) No immunodeficiencies No metabolic disease No social situation that would interfere with follow up Not pregnant Negative pregnancy test

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 1999-05

CONTACTS AND LOCATIONS:
Overall Officials: Frank T. Gentile, Study Chair — Curis, Inc.